CLINICAL TRIAL: NCT01366105
Title: Use of Negative Pressure Wound Therapy for At Risk Surgical Closures
Brief Title: VAC NPWT KCI Dressing Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christopher Attinger, M.D., Chief of the Division of the Center for Wound Healing, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-293
Record Dates: First submitted 2011-05-26; First posted 2011-06-03 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Surgical Wound Infection
Keywords: Wound healing; Negative Pressure Wound Therapy; V.A.C.; Incision
MeSH Terms: conditions — Surgical Wound Infection; Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Dressing (No Intervention): Incisions that were dressed with a sterile dry dressing at end of operation.
- Negative Pressure Wound Therapy (Experimental): Incisions dressed with a V.A.C. (NPWT) postoperatively.
  Interventions: Device: V.A.C. by K.C.I.

INTERVENTIONS:
Device: V.A.C. by K.C.I. — Negative Pressure Wound Therapy, Delivered by Vacuum Assisted Closure (KCI) across closed surgical incision at completion of surgery
  Other Names: V.A.C. (Kinetic Concepts Incorporate)
  Arms: Negative Pressure Wound Therapy

SUMMARY:
In this study, the investigators propose using negative pressure wound therapy (NPWT) to aid in wound healing along the lines of closure for lower extremity amputation and complex abdominal wounds. This study is designed to be a prospective, randomized clinical trial to evaluate the effectiveness of NPWT versus accepted standard surgical dressings on these wounds. Study participants will be randomized to one of the two treatment groups (NPWT vs. standard dressing) prior to surgery, and will be followed in the post operative period to monitor the effects on their surgical closures. The experimental group will consist of participants receiving NPWT and will have a Vacuum Assisted Closure (V.A.C., KCI inc.) device placed intra-op along the line of closure. The control group will receive a standard surgical dry sterile dressing. The surgical closures will be assessed after three days of treatment as well as the first outpatient post-op visit and any subsequent visits through the following 6 months. By doing so, the investigators hope to demonstrate the utility of NPWT on difficult, at risk surgical closures. Additionally, the investigators hope to show a difference in clinical outcome of incisions treated by NPWT over our current standard technique.

All patients in the principal and co-investigators practice who are scheduled to undergo lower extremity amputation or complex abdominal closure will be eligible for enrollment in this prospective randomized study. There are no exclusion criteria. Informed consent will be obtained pre-operatively. Data collection will include basic demographic data, disease history, past medical and social history as well key data relating to wound healing (infection, wound dehiscence or breakdown) and hospital course (length of stay, operative complications). The investigators will use simple statistical methods (ANOVA and chi-squared analysis) to compare surgical wound healing between the two populations. The only deviation from current standard of care in these populations includes utilizing a V.A.C. system on the closure line of the experimental group versus the standard dry sterile dressing.

DETAILED DESCRIPTION:
No further description is desired

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to wound center undergoing wound treatment with expected closure of wounds including: Midfoot amputations, below knee amputations, knee disarticulations, above knee amputations, and trunk wounds
* wounds must be closed primarily without the use of grafts

Exclusion Criteria:

* any patient <18 years old
* any patient whose wound is unable to be closed primarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incisional Dehiscence | last post operative visit, up to 2 years
  any amount of incisional dehiscence noted post-operatively
Post operative infection | last post operative visit, up to 2 years
  Post operative infection as noted by increased white count, clinical findings supporting infection (erythema, purulence, wound drainage)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Attinger, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Masden D, Goldstein J, Endara M, Xu K, Steinberg J, Attinger C. Negative pressure wound therapy for at-risk surgical closures in patients with multiple comorbidities: a prospective randomized controlled study. Ann Surg. 2012 Jun;255(6):1043-7. doi: 10.1097/SLA.0b013e3182501bae. PMID 22549748